CLINICAL TRIAL: NCT04684264
Title: Transforming the Primary Prevention Paradigm for Heart Failure: Feasibility of the Implementation of Tools for Heart Failure Risk Prediction
Brief Title: Feasibility of the Implementation of Tools for Heart Failure Risk Prediction
Acronym: FIT-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Sadiya Khan, Assistant Professor of Medicine (Cardiology) and Preventive Medicine (Epidemiology), Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU00210780
Record Dates: First submitted 2020-12-11; First posted 2020-12-24 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure; Cardiovascular Risk Factor
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist-directed collaborative practice (Experimental): Participants will be referred to a pharmacist-directed collaborative practice for heart failure prevention.
  Interventions: Other: Heart Failure Prevention Clinic
- Usual care (No Intervention): Participants will receive usual care with their primary care physician.

INTERVENTIONS:
Other: Heart Failure Prevention Clinic — Heart Failure Prevention Clinic is a pharmacist-directed practice in collaboration with an attending cardiologist that uses evidence-based guidelines to optimize medications and lifestyle interventions for heart failure prevention.
  Arms: Pharmacist-directed collaborative practice

SUMMARY:
The purpose of this study is to gather information to develop a heart failure screening and prevention program.

DETAILED DESCRIPTION:
All participants will undergo phlebotomy for specimen collection (BNP, hs-cTn, BMP and lipid testing, biorepository storage) and baseline echocardiography. All participants will additionally be administered a health and lifestyle questionnaire, undergo measurement of vital signs, and receive uniform education on heart-healthy lifestyle and signs and symptoms of heart failure. Participants who are randomized to the intervention arm will receive a referral to Heart Failure Prevention Clinic, a pharmacist-directed practice in collaboration with an attending cardiologist, where they will be followed for 1 year, with their primary care physician updated after each visit. The information from their BNP, hs-cTn, and echocardiography will be provided to them and their primary care physicians as well as the pharmacist and cardiologist team members. The participants (and their primary care providers) who are randomized to usual care will be blinded to their BNP and hs-cTn values and echocardiography results.

ELIGIBILITY:
Inclusion Criteria:

* 10-year risk of heart failure >5% based on the PCP-HF equations
* At least one primary care visit in the last 12 months
* At least one additional primary care visit in the last 5 years
* Had cholesterol and glucose checked within the past 5 years

Exclusion Criteria:

* History of cardiovascular disease
* Signs and symptoms of heart failure
* Estimated glomerular filtration rate <45 mL/min/1.73m^2
* Stage 3 or 4 cancer
* Pregnancy

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in BNP at 1 year | baseline, 1-year
  All participants will have brain natriuretic peptide (BNP) measured at baseline and at 1-year follow-up.

SECONDARY OUTCOMES:
Change from baseline in hs-cTn at 1 year | baseline, 1-year
  All participants will have high sensitivity cardiac troponin (hs-cTn) measured at baseline and at 1-year follow-up.
Change from baseline in BP at 1 year | baseline, 1-year
  All participants will have systolic blood pressure and diastolic blood pressure measured at baseline and at 1-year follow-up.
Change from baseline in weight status at 1 year | baseline, 1-year
  All participants will have weight and BMI measured at baseline and at 1-year follow-up.
Change from baseline in serum glucose at 1 year | baseline, 1-year
  All participants will have serum glucose measured at baseline and at 1-year follow-up.
Change from baseline in LDL at 1 year | baseline, 1-year
  All participants will have LDL cholesterol measured at baseline and at 1-year follow-up.
Change from baseline in estimated glomerular filtration rate at 1 year | baseline, 1-year
  All participants will have estimated glomerular filtration rate measured at baseline and at 1-year follow-up.
Change from baseline in creatinine at 1 year | baseline, 1-year
  All participants will have creatinine measured at baseline and at 1-year follow-up.
Smoking quit attempt or cessation | baseline, 1-year
  All participants will be asked about smoking status at baseline and at 1-year follow-up. Outcome is, among patients who were current smokers at baseline, quit attempt or no smoking at 1 year.

OTHER OUTCOMES:
Medication adherence at 1 year | 1 year
  All participants will be asked about adherence to medications (if applicable) using questions of nonadherence from the Atherosclerosis Risk in Communities study.
Change from baseline in E/e' ratio at 1 year | baseline, 1-year
  All participants will undergo echocardiogram at baseline and at 1 year.
Change from baseline in left ventricular mass index at 1 year | baseline, 1-year
  All participants will undergo echocardiogram at baseline and at 1 year.
Biomarker assay | baseline
  All participants will have biorepository storage of serum and plasma at baseline. An exploratory analysis will use a commercial biomarker array to investigate correlations with echocardiogram, BNP, and hs-cTn results.
Change from baseline in fruit and vegetable intake | baseline, 1-year
  All participants will be asked about fruit and vegetable intake at baseline and at 1 year. Outcome will be measured in servings/week.
Change from baseline in salt intake | baseline, 1-year
  All participants will be asked about salt intake at baseline and at 1 year using a 5-point Likert scale (always, often, sometimes, rarely, never). A higher score on this scale is preferable.
Change from baseline in physical activity | baseline, 1-year
  All participants will be asked about physical activity at baseline and at 1 year. Outcome is measured in minutes of moderate-intensity activity per week. Vigorous-intensity activity will count as twice the equivalent duration of moderate-intensity activity.
Change from baseline in sedentary behavior | baseline, 1-year
  All participants will be asked about sedentary behavior at baseline and at 1 year. Outcome is measured in minutes of sedentary behavior per day.
Change from baseline in health utility | baseline, 1-year
  Health utility will be measured by the EurolQol 5 Dimensions 5 Levels (EQ-5D-5L) instrument. Typical scores range from 0 to 1, with 1 being ideal health-related quality of life.
Change from baseline in overall health | baseline, 1-year
  Overall health will be measured by the EurolQol Visual Analog Scale (EQ VAS) instrument. Scores range from 0-100, with 100 being the highest overall health.

CONTACTS AND LOCATIONS:
Overall Officials: Sadiya Khan, MD, MSc, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Preventive Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang MC, Dolan B, Huang X, Freaney PM, Freed BH, Vega L, Markoski N, Wainright A, Kane B, Seegmiller LE, Shah SJ, Yancy CW, Neeland IJ, Ning H, Lloyd-Jones DM, Khan SS. Feasibility of the Implementation of Tools for Heart Failure Risk Prediction: A Randomized Controlled Pilot Trial. JACC Adv. 2025 Aug;4(8):102004. doi: 10.1016/j.jacadv.2025.102004. Epub 2025 Jul 14. PMID 40664007
- [Derived] Wang MC, Dolan B, Freed BH, Vega L, Markoski N, Wainright AE, Kane B, Seegmiller LE, Harrington K, Lewis AA, Shah SJ, Yancy CW, Neeland IJ, Ning H, Lloyd-Jones DM, Khan SS. Rationale and Design of a Pharmacist-led Intervention for the Risk-Based Prevention of Heart Failure: The FIT-HF Pilot Study. Front Cardiovasc Med. 2021 Nov 29;8:785109. doi: 10.3389/fcvm.2021.785109. eCollection 2021. PMID 34912869